CLINICAL TRIAL: NCT00638573
Title: The Incretin Effect in Patients With Chronic Pancreatitis With and Without Secondary Diabetes Mellitus
Brief Title: The Incretin Effect in Patients With Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Filip K. Knop, Diabetes Research Division, Department of Internal Medicine F, Gentofte Hospital, University of Copenhagen
Other Study IDs: KA04034
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2008-03

CONDITIONS: Chronic Pancreatitis; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Pancreatitis, Chronic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The phenomenon that oral glucose elicits a higher insulin response than does intravenous (iv) glucose, even at identical plasma glucose (PG) profiles (isoglycemia), is called the incretin effect. In type 2 diabetes mellitus (T2DM) the incretin effect has been shown to be markedly reduced or even abolished. It is not known whether the reduced incretin effect in T2DM is a primary event leading to T2DM or if it is merely a consequence of the diabetic state. To answer this question the investigators plan to estimate the incretin effect in 8 patients with secondary diabetes mellitus (DM) to chronic pancreatitis (CP) and compare it to the incretin effect of 8 patients with CP and normal glucose tolerance (NGT). Eight patients with T2DM and 8 healthy control subjects are studied for comparison. The incretin effect is measured by a 50-g oral glucose tolerance test and an isoglycemic intravenous glucose infusion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pancreatitis with secondary diabetes mellitus
* Diagnosis of chronic pancreatitis with normal glucose tolerance
* Diagnosis of type 2 diabetes
* Normal level of hemoglobin
* Normal level of se-creatinine

Exclusion Criteria:

* GAD-65 autoantibodies
* ICA autoantibodies
* Albuminuria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pancreatitis with and without secondary diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2006-01; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, Principal Investigator — University of Copenhagen; Jens J Holst, MD DMSc, Study Director — University of Copenhagen; Thure Krarup, MD DMSc, Study Director — Gentofte University Hospital
Locations (1):
- Gentofte University Hospital, Hellerup, Copenhagen County, Denmark